CLINICAL TRIAL: NCT00507208
Title: Dynasplint Therapy for Trismus in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Dynasplint Systems, Inc. (Industry)
Responsible Party: Principal Investigator, William Carroll, MD, Professor of Otolaryngology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F070323014; HNO 0602 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Trismus
Keywords: trismus; head and neck cancer
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynasplint (Experimental): Participants randomized to this arm will be treated with the Dynasplint Trismus System
  Interventions: Device: Dynasplint Trismus System
- Control (Active Comparator): Participants randomized to this arm will use tongue depressors for 3 months and if there is no improvement in their mouth opening at this timepoint, they will crossover to the Dynasplint Trismus System
  Interventions: Other: Tongue Depressors

INTERVENTIONS:
Device: Dynasplint Trismus System — The Dynasplint System will be used for 6 months.
  Arms: Dynasplint
Other: Tongue Depressors — Tongue depressors to be used for 3 months at which time mouth opening will be measured. If there is no change then the patient will crossover to the Dynasplint Trismus System for another 3 months.
  Arms: Control

SUMMARY:
The purpose of this study is to compare the use of the Dynasplint Trismus System to routine trismus treatment in improving the ability of opening the mouth in a randomized trial. This study will also determine what effects, good and/or bad, this procedure has on the participant. Participants will be randomly assigned to the Dynasplint Trismus System or to routine treatment with tongue depressors.

DETAILED DESCRIPTION:
This trial is a single-institution, randomized study to evaluate the effectiveness of the Dynasplint Trismus System (DTS) for patients with trismus. Improvement of mouth opening and quality of life of participants using DTS will be compared to improvement of mouth opening and quality of life of participants using standard therapy. Standard therapy will be the use of tongue depressors. Crossover from standard therapy to DTS will be implemented if at three months there is no improvement in mouth opening when using tongue depressors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with <= 30mm mouth opening who have undergone treatment for head and neck cancer. (If the patient is edentulous then mouth opening must be <= 40mm.)
2. Patients who are receiving or have completed treatment for head and neck cancer (surgery, radiation, chemotherapy alone or in any combination).
3. Patients must be completely recovered from any radiation induced oral mucositis.
4. Age =>19 years.
5. Patients must sign informed consent.

Exclusion Criteria:

1. Severe periodontal or gum disease that has caused teeth to be loose.
2. Any systemic disease that causes blistering of the oral mucosa.
3. Any condition that renders the patient unable to understand the informed consent.
4. Participants who are not able to comply with protocol activities.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carroll, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Otolaryngology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants randomized to this arm will use tongue depressors for 3 months and if there is no improvement in their mouth opening at this timepoint, they will crossover to the Dynasplint Trismus System for 3 months.
Period: Overall Study
Arm/Group | Dynasplint | Control
Started | 27 | 26
Received Dynasplint in Crossover | 0 | 3
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynasplint | Control | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 18 | 20 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 17 | 40
  African-American | 3 | 9 | 12
  Hispanic | 1 | 0 | 1
Prior Treatment [Number; unit: participants] — Type of treatment completed prior to enrollment in the study
  participants
    Chemoradiation & Surgery | 23 | 22 | 45
    Surgery only | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Improved MIO Using Either the Dynapslint System or Tongue Depressors
Description: Number of participants who demonstrated improved maximal incisial opening (MIO), the distance from the tips of the upper and lower incisors on maximal effort. Successful improvement is defined as > 5mm improvement from the baseline measurement.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Dynasplint | Control
Number analyzed (Participants) | 27 | 26
participants
  MIO improvement > 5mm or more | 12 | 12
  MIO improvement < 5 mm or less | 7 | 7
  unknown MIO improvement | 8 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dynasplint | Control
Serious Adverse Events (participants affected / at risk) | 11/27 | 6/26
Other Adverse Events (participants affected / at risk) | 9/27 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dynasplint (N=27) | Control (N=26)
oral fistula (Gastrointestinal disorders) | 1 | 0
esophageal stenosis (Gastrointestinal disorders) | 1 | 1
upper GI bleed (Gastrointestinal disorders) | 1 | 0
facial cellulitis (Infections and infestations) | 1 | 0
injury to carotid artery (Injury, poisoning and procedural complications) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
debulking of scar tissue (Surgical and medical procedures) | 1 | 0
mandibular debridement (Surgical and medical procedures) | 1 | 0
disease recurrence resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
planned procedures prior to radiation tx (Surgical and medical procedures) | 0 | 1
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dynasplint (N=27) | Control (N=26)
oral pain (Gastrointestinal disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes